CLINICAL TRIAL: NCT02048228
Title: Study of Clopidogrel and Ticagrelor Anti-Platelet Treatment Using an Individualized Strategy Based on Genotyping in Chinese ACS Patients
Brief Title: Genotyping Guided Individualized Treatment of Clopidogrel and Ticagrelor in ACS
Acronym: GI-CT
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Tong Yin, MD, PhD, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCT01417884
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2014-04-11 (Estimated); Status verified 2014-04

CONDITIONS: CLOPIDOGREL, POOR METABOLISM of (Disorder)
Keywords: Clopidogrel,; Pharmacogenetics,; Platelet reactivity,; CYP2C19,; point-of-care
MeSH Terms: interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- genotyping guided therapy (Experimental): Patients randomized to the genotyping guided therapy arm will have their CYP2C19*2 carrier status determined at the time before antiplatelet therapy with subsequent alteration in antiplatelet therapy for *2 carriers.CYP2C19*2 carriers will be given 90 mg ticagrelor twice daily, and non-carriers will be given 75 mg clopidogrel daily.
  Interventions: Drug: genotyping guided therapy Ticagrelor, Clopidogrel
- Standard Therapy (Active Comparator): Patients randomized to the Standard Therapy arm will not undergo genotyping. All patients will be administrated with clopidogrel 75 mg daily for 5 consecutive days.
  Interventions: Drug: standard therapy clopidogrel

INTERVENTIONS:
Drug: genotyping guided therapy Ticagrelor, Clopidogrel — CYP2C19*2 carriers will be given 90 mg ticagrelor twice daily, and non-carriers and patients in the standard treatment group will be given 75 mg clopidogrel daily.
  Other Names: Ticagrelor; Clopidogrel
  Arms: genotyping guided therapy
Drug: standard therapy clopidogrel — All patients will be administrated with clopidogrel 75 mg daily for 5 consecutive days.
  Other Names: clopidogrel
  Arms: Standard Therapy

SUMMARY:
Clopidogrel, in addition to aspirin, is the cornerstone of therapy in patients suffering from Acute coronary syndrome. However, the platelet inhibitory response to clopidogrel varies substantially among individuals. Several loss-of-function polymorphisms have been identified that may influence clinical outcome in patients presenting with acute coronary syndromes (ACS) who are treated with clopidogrel. However their contribution to high on-treatment platelet reactivity (HPR) in clopidogrel treated Chinese patients is less known. As far as we know, ticagrelor is not dependent on gene-based metabolic activation and demonstrated greater clinical efficacy than clopidogrel in a recent secondary prevention trial. we will conduct an interventional study to compare the antiplatelet efficiency between clopidogrel and ticagrelor by the guidance of CYP450 2C19*2 (CYP2C19*2) , using Taqman genotyping method.

DETAILED DESCRIPTION:
Clopidogrel, in addition to aspirin, is the cornerstone of therapy in patients suffering from Acute coronary syndrome. However, the platelet inhibitory response to clopidogrel varies substantially among individuals. Several loss-of-function polymorphisms have been identified that may influence clinical outcome in patients presenting with acute coronary syndromes (ACS) who are treated with clopidogrel.

Mounting evidence suggests a crucial role for the loss-of-function CYP2C19*2 genetic variant. Carriers of CYP2C19*2 allele were at 30% higher risk for major adverse clinical events compared to non-carriers. CYP2C19*2 alone was also associated with increased mortality and stent thrombosis. These findings led the American Food and Drug Administration to issue a boxed warning for clopidogrel stating that poor metabolizers may not receive the full benefit of the drug. Thus, routine genotyping in the context of dual anti-platelet therapy is necessary.

Individual dual anti-platelet treatment is feasible to give the presence of treatment alternatives such as ticagrelor that is not dependent on gene-based metabolic activation and demonstrated greater clinical efficacy than clopidogrel. Individualized administration of ticagrelor may have the potential to successfully minimize adverse ischemic events.

200 patients undergoing percutaneous coronary intervention (PCI) for treatment of non-ST-elevation acute coronary syndrome or stable coronary artery disease will be eligible for enrollment. Patients will be randomly assigned to a strategy of genotyping(using Taqman genotyping method) or standard treatment . CYP2C19*2 carriers will be given 90 mg ticagrelor twice daily, and non-carriers and patients in the standard treatment group will be given 75 mg clopidogrel daily. At the end of the 5 day antiplatelet treatment, efficacy of the treatment strategies will be evaluated using light transmittance aggregometry (LTA) method.

ELIGIBILITY:
Inclusion Criteria:

The diagnosis of ACS including unstable angina (UA),non-ST elevation myocardial infarction(NSTEMI),and ST-elevation MI (STEMI) is according to the American Heart Association/American College of Cardiology (AHA/ACC) criteria

Exclusion Criteria:

known contraindication to dual anti-platelet therapy, history of chronic inflammatory disease, steroidal and non-steroidal anti-inflammatory drugs use, previous administration of antiplatelet drugs within 1 month before coronary artery angiography, illicit drug abuse, significant bleeding, cerebrovascular event within 3months, and/or major surgery within 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-03 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Clopidogrel response status as measured by the LTA assay in CYP2C19*2 carriers. | Day 5 of enrollment
  The primary endpoint is the proportion of CYP2C19*2 carriers with a platelet aggregation more than 59% after 5 days of antiplatelet therapy.The deﬁnition of high on-treatment platelet reactivity is derived from previous studies that had identiﬁed platelet aggregation more than 59% as optimum cutoff values for prediction of increased risk of major adverse cardiovascular events in Chinese patients.

CONTACTS AND LOCATIONS:
Overall Officials: Tong Yin, MD, PhD, Principal Investigator — Institute of Geriatric Cardiology, General Hospital of Chinese People's Liberation
Locations (1):
- General Hospital of Chinese People's Liberation Army, Beijing, China